CLINICAL TRIAL: NCT05210361
Title: Critical Windows in the Development of Asthma Endotypes and Phenotypes in High-Risk Toddlers
Acronym: WINDOWS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-3116; U01AI160033 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-01-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Asthma in Children; Wheezing
Keywords: childhood asthma; recurrent wheeze; asthma phenotypes; asthma endotypes; asthma development
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn more about how asthma develops in early childhood. This will help doctors understand how to prevent and treat asthma better.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 months to 36 months at first research encounter
* For enrollment in Emergency Department (ED)/Inpatient Visit: Presentation to the ED/Inpatient with an acute wheezing episode AND either evidence of at least one prior wheezing episode documented in the electronic medical record (i.e., wheezing, pneumonitis, bronchiolitis, reactive airways disease, or asthma) that occurred ≥ 14 days from current episode, or caregiver report of one of the following:

  * Child has had wheezing or whistling in the chest at any time in the past lasting at least 24 hours and occurring at least 14 days prior to the current ED visit
  * Child has been treated with albuterol or used an inhaler or a nebulizer at least 14 days prior to the current ED visit
  * Caregiver has been told that their child has bronchiolitis, asthma, or reactive airways disease at least 14 days prior to the current ED visit
* For enrollment in Visit 1: At least three separate wheezing episodes, separated by at least 14 consecutive days without a wheezing episode (wheezing lasting ≥ 24 hours), as reported by parent/caregiver or patient's care provider and/or documented in the patient's medical record

  * Third episode may be at time of presentation to ED or admission as inpatient (IP) to hospital when recruitment would occur (Visit ED/IP)
  * Bronchiolitis and wheezing/asthma exacerbations are considered wheezing episodes
  * The wheezing episode does not require treatment with bronchodilators
* Live within a US Office of Management and Budget-defined Metropolitan Statistical Area (MSA) and meet at least one of these criteria:

  1. Have publicly funded health insurance AND/OR
  2. Live in a census tract within an MSA where ≥10% of families have income below the poverty level

Exclusion Criteria:

* Wheeze attributed to alternative diagnoses other than bronchiolitis or asthma, including congenital anatomical abnormalities, foreign body aspiration, chronic lung disease of prematurity, other chronic lung disorders such as cystic fibrosis, and cardiac, immune, and gastrointestinal disorders.
* Gestational age < 32 weeks.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of toddlers at high risk for developing childhood asthma, living in low-income urban communities in the Denver Metropolitan Area in Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of persistent asthma | At visit 5, after 4 years of participation in the longitudinal study
  Children will be classified as having persistent asthma if at least 1 of the following 3 conditions are met:
  1. Doctor Diagnosis: a parent-reported physician's diagnosis of asthma between age 4 and 7 years plus asthma symptoms or the use of asthma controller medication for at least 6 of the past 12 months
  2. Lung Function: bronchodilator-induced improvement of forced expiratory volume in 1 second (FEV1) by 10% or more plus asthma symptoms or use of asthma controller medication for at least 6 of the past 12 months
  3. Symptoms: report in the past 12 months of 2 or more wheezing episodes, 2 or more doctor's office visits for asthma/wheeze, 1 or more hospitalizations for asthma/wheeze, or use of controller medications for at least 6 of the past 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Liu, MD, Principal Investigator — University of Colorado, Denver; Katharine Hamlington Smith, PhD, Study Director — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States